CLINICAL TRIAL: NCT04150926
Title: The Effect of Black Currant on Postprandial Glucose Metabolism
Acronym: MAQUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Savonia University of Applied Sciences (Other); Regional Development Company SavoGrow (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 894/2019
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Postprandial Hyperglycemia; Prediabetic State
Keywords: berries; black currant; glucose; glycemia; quinoa
MeSH Terms: conditions — Hyperglycemia; Prediabetic State | interventions — black currant oil

STUDY DESIGN:
Intervention Model Description: Meal studies in randomised order
Who Masked: Participant
Masking Description: Products are visibly differing from each other.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Black currant puree (Experimental): Black currant puree
  Interventions: Other: Black currant
- Black currant-quinoa product (Active Comparator): Black currant-quinoa product
  Interventions: Other: Black currant-quinoa product
- Quinoa base (Active Comparator): Quinoa base is used for the black currant-quinoa product.
  Interventions: Other: Quinoa base
- Liquid with glucose, fructose and sucrose (No Intervention): Liquid with glucose, fructose and sucrose

INTERVENTIONS:
Other: Black currant — The effect of black currant puree will be compared with black currant-quinoa product, quinoa base and with liquid with glucose, fructose and sucrose
  Experimental: Black currant and quinoa product
  Active Comparator: Quinoa base Meal study comparing the effect of black currant puree with liquid with glucose, fructose and sucrose, black currant and quinoa product and quinoa base
  Arms: Black currant puree
Other: Black currant-quinoa product — The effect of black currant puree will be compared with black currant-quinoa product
  Arms: Black currant-quinoa product
Other: Quinoa base — The effect of black currant puree will be compared with quinoa base
  Arms: Quinoa base

SUMMARY:
The study examines the effect of black currant on glucose and insulin concentrations after a meal. In addition, the cytokine and free fatty acids levels are of interest.

DETAILED DESCRIPTION:
The study examines the effect of black currant on glucose and insulin concentrations after a meal.

Healthy (n= 30) volunteers are recruited to participate in four consecutive visits in the research laboratory, when four meals are served in randomised order. Meals are: black currant puree, black currant and quinoa based snack, quinoa base and liquid containing glucose, fructose and sucrose. The meals contain the same amount of carbohydrates.

In addition to glucose and insulin concentration, cytokine and free fatty acid concentrations are measured after each meal.

ELIGIBILITY:
Inclusion Criteria:

* age: 25-65 years
* BMI: 20-28 kg/m2
* Perceived health status: Good

Exclusion Criteria:

* fasting glucose: > 7.0 mmol/l
* LDL-cholesterol: > 3.0 mmol/l
* total cholesterol: > 6.5 mmol/l
* blood pressure : > 160/100 mmHg
* weight change of > 5% during previous 6 months or active weightreduction
* no serious chronic diseases
* one exception of the exclusion criteria maybe accepted after the MD consideration

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose concentration | 0 minutes until 180 minutes
  Glucose concentration after meal
Insulin concentration | 0 minutes until 180 minutes
  Insulin concentration after meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No
Anonymised data maybe shared in the future.